CLINICAL TRIAL: NCT01159652
Title: Hypnotic Medications and Sleep-dependent Memory Consolidation: the Effect of Variable Drug Exposure During the Night
Brief Title: Hypnotic Medications and Memory: Effect of Drug Exposure During the Night
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's Hospital, Chesterfield, Missouri (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 63-SR-10
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Sleep; Memory
Keywords: sleep; memory; hypnotics; zaleplon; zolpidem; Sonata; Ambien; Hypnotics and Sedatives; Polysomnography; Monitoring, sleep
MeSH Terms: interventions — zaleplon; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bedtime Placebo (Placebo Comparator)
  Interventions: Drug: bedtime placebo
- Middle of the Night Placebo (Placebo Comparator)
  Interventions: Drug: middle of the night placebo
- Zolpidem (Experimental)
  Interventions: Drug: zolpidem extended release
- Zaleplon (Experimental)
  Interventions: Drug: zaleplon

INTERVENTIONS:
Drug: zaleplon — 10 mg
  Other Names: Sonata
  Arms: Zaleplon
Drug: zolpidem extended release — 12.5 mg
  Other Names: Ambien CR
  Arms: Zolpidem
Drug: bedtime placebo — placebo
  Arms: Bedtime Placebo
Drug: middle of the night placebo — placebo
  Arms: Middle of the Night Placebo

SUMMARY:
The purpose of this study is to determine the effect of two hypnotic medications, zolpidem extended release and zaleplon, on memory. It is expected that a hypnotic with shorter drug duration will allow greater memory consolidation than a hypnotic with longer drug duration.

DETAILED DESCRIPTION:
A growing body of evidence has demonstrated that sleep promotes memory consolidation in healthy individuals. However, little research has been conducted regarding the effect of hypnotics on sleep-dependent memory. One study found that zopiclone (7.5 mg), but not brotizolam (0.25 mg), impaired sleep-dependent memory consolidation in normal sleepers. Another study reported significant impairment of sleep-dependent memory on a motor task with triazolam (0.375 mg), but not with zolpidem immediate release (10 mg). These studies provide some evidence that sedative-hypnotic drugs may impair sleep-dependent memory consolidation, but further investigation is clearly needed in this area. Because hypnotics are commonly prescribed for insomnia, it is important to determine if there is a significant risk of impairment in sleep-dependent memory consolidation associated with these medications. Further, investigation of alternative doses and drug regimens upon memory consolidation appears warranted.

The purpose of the current study is to determine the effect of two hypnotic medications on sleep-dependent memory consolidation in normal sleepers. Zolpidem extended release, which will be active for most of the sleep period when administered at bedtime, will be compared to zaleplon, which will be active for half of the sleep period when administered in the middle of the night. This comparison allows us to address the question of whether a few hours of drug-free sleep results in better memory consolidation than sleep with drug throughout the night.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age
* no sleep complaints or problems
* good sleep quality per questionnaire
* sufficient time in bed each night

Exclusion Criteria:

* any clinically significant unstable medical condition
* recent psychiatric disorder
* prior diagnosis or symptoms of a sleep disorder
* recent history of substance abuse
* recent use of prescription hypnotic medication or over-the-counter sleep aid
* recent use of psychotropic medication
* history of adverse reaction to benzodiazepines
* body mass index > 36
* currently pregnant or nursing
* currently working rotating or night shift
* consumption of > 700 mg per day of xanthine-containing food or beverages
* consumption of > 14 units of alcohol per week
* smoke > 1 pack of cigarettes per day, use of chewing tobacco more than 3 times per day, or unable to refrain from smoking or chewing without distress or discomfort while in the sleep laboratory

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Memory | 8 timepoints: 4 evenings and 4 mornings
  Two memory tasks will be used to assess memory.

CONTACTS AND LOCATIONS:
Overall Officials: Janine M Hall-Porter, PhD, Principal Investigator — St. Luke's Hospital
Locations (1):
- St. Luke's Hospital Sleep Medicine and Research Center, Chesterfield, Missouri, United States

REFERENCES:
- [Background] Greenblatt DJ, Harmatz JS, von Moltke LL, Ehrenberg BL, Harrel L, Corbett K, Counihan M, Graf JA, Darwish M, Mertzanis P, Martin PT, Cevallos WH, Shader RI. Comparative kinetics and dynamics of zaleplon, zolpidem, and placebo. Clin Pharmacol Ther. 1998 Nov;64(5):553-61. doi: 10.1016/S0009-9236(98)90139-4. PMID 9834048
- [Background] Weinling E, McDougall S, Andre F, Bianchetti G, Dubruc C. Pharmacokinetic profile of a new modified release formulation of zolpidem designed to improve sleep maintenance. Fundam Clin Pharmacol. 2006 Aug;20(4):397-403. doi: 10.1111/j.1472-8206.2006.00415.x. PMID 16867025